CLINICAL TRIAL: NCT06208111
Title: A Clinical Trial of Cognitive Behavior Therapy for Depression, Stigmatization, Excessive Worries, and Emotional Management Among Women Facing Partner Violence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Qasir Abbas, Dr.Qasir Abbas Assistant Professor Clinical Psychology, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GovernmentGUF
Record Dates: First submitted 2023-11-29; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cognitive Behaviour Therapy
Keywords: Depression Worries Stigma Emotion Cognitive behavior therapy
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A randomized control trial design will be used in this study. it would be two arm study and there would be two groups an experimental and a waitlist control group. The experimental group will receive intervention and another group will be placed on the waitlist. in this research parallel group design would be used. we will give treatment to all participants in a parallel way. The allocation ratio and framework would be equivalency i.e, the treatment group and control group be equal number of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Experimental Group:
  participants in the experimental group would receive 8-10 Cognitive Behaviour Therapy-based therapeutic sessions.
  Interventions: Behavioral: cognitive behavioral therapy
- control group (No Intervention): Participants in the control group did not receive the said Cognative Behaviour Therapy intervention

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — cognitive behavioral therapy would be used as intervention strategy for women facing partner violence to Clear about actual problems, re-educate about the issue of domestic problems and mental health, Logical expectations, Identify negative automatic thoughts,Thinking errors, and Improve understanding to identify which stressors trigger negative emotions. Moreover, this intervention will help to Prepare women how to deal with stress and overcome the reaction.
  Arms: Treatment group

SUMMARY:
1. Aim to investigate the effectiveness of Cognitive Behavior Therapy for Depression, Stigmatization, Excessive Worries, and Emotional Management among Women Facing Partner Violence
2. To explore the effectiveness of CBT in managing depressive symptoms, stigma, worries, and emotional disturbance among women facing partner violence.

DETAILED DESCRIPTION:
In this Randomized control trial, N=180 participants would be enrolled for eligibility assessment from different shelter homes in the cities of Punjab after the eligibility assessment and screening 108 participants would be allocated to experimental and waitlist treatment conditions. Participants will be allocated through matchable group characteristics. Participant's age range would be between 18 to 45 years. Each of the group will be comprised of the same number of participants. Both groups will be pre-tested and results will be recorded. A cognitive behavior therapy-based treatment plan will be formulated to address Depression, Stigmatization, Excessive Worries, and Emotional Management among Women Facing Partner Violence. 8-10 CBT-based therapeutic sessions with 60 minutes will be conducted with the participant in a one-on-one setting.

ELIGIBILITY:
Inclusion Criteria:

* Women living in the institutions for at least 2 weeks because of partner violence
* Second eligibility criteria would be women with a minimum of 1 year of marital relationship will be included.
* The age range would be 18 -48 years.
* Women whose scores are above average on the partner violence scale would be included in the study

Exclusion Criteria:

* Women greater than 48 years and less than 18 years will be excluded.
* Women with medical and psychiatric comorbidities will be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Eligibility Assessment: | 2-4 weeks
  Initially, we enroll the women for eligibility assessment. Women who live in shelter home will be part of the study. After choosing, the Participants demographic form will be filled out. In demographic form information related to age, marital status, marriage type, family system, children, education and financial status. After this, eligible participants will be referred for psychological evolution.
Depression: | after allocation 1 week
  Depression will be assessed by using Depression Anxiety Stress Scale. A score of 13, 20, 27 9, 14, 19, 18, 25, 33 corresponding to the categorization of mild moderate and sever level of depression, anxiety and stress respectively.
Stigmatization: | after allocation 1 week
  Intimate Partner Violence Stigma Scale will asses stigmatization. Higher score will indicate high-level stigma whereas low score indicate low level of stigma.
Excessive Worries: | after allocation 1 week
  Excessive worries will be assessed by using Generalized Anxiety Scale GAD-7. A score of 4,9,15 corresponding to the categorization of mild moderate and sever level of worries. Score greater than 15 will show the severe level of Anxiety.
Emotional Management: | after allocation 1 week
  Emotional Management will be assessed by using Emotional Regulation Scale. This scale comprised of ten items. Higher score on items 1,3,5,7,8,10 will show the higher level of Cognitive Reappraisal and higher score on items 2, 4, 6, and 9 will show the higher level of Expressive Suppression. Low score on these items will show the lower level of Cognitive Reappraisal and Expressive Suppression.
Partner Violence: | after allocation 1 week
  Karachi Domestic violence scale will be used to assess the intimate partner violence. The lowest score on KDVSS will be 0 and highest score on this scale will be 105.The cut-off score for indication that person facing the domestic abuse will be <29.

SECONDARY OUTCOMES:
Duration of illness | at the time of pre assessment (1week)
  They will be assessed through interview information
HISTORY Of Domestic violence | after allocation at pre assessment (1week)
  they will be assessed through history taking information

CONTACTS AND LOCATIONS:
Overall Officials: Qasir Abbas, PHD, Principal Investigator — Government College University Faisalabad
Locations (1):
- Qasir Abbas, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No